CLINICAL TRIAL: NCT01659099
Title: Randomized Phase III Study Using a Pet-driven Strategy and Comparing GA101 OR Rituximab Associated to a Chemotherapy Delivered Every 14 Days (ACVBP or CHOP) in DLBCL CD20+ Lymphoma Untreated Patients From 18 to 60 Presenting With 1 or More Adverse Prognostic Factors of the Age-adjusted IPI
Brief Title: GA In NEwly Diagnosed Diffuse Large B Cell Lymphoma
Acronym: GAINED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: experimental treatment not Superior to standard - no need to continue the follow-up
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAINED
Record Dates: First submitted 2012-07-04; First posted 2012-08-07 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Diffuse Large B Cell Lymphoma CD20 Positive
Keywords: DLBCL; aa-IPI > or equal to 1; Diagnosis; 18 to 60 years; Lymphoma
MeSH Terms: conditions — Disease; Lymphoma | interventions — obinutuzumab; Rituximab; Doxorubicin; Cyclophosphamide; Prednisone; Bleomycin; Vindesine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GA101 (Experimental): GA101 - Chemotherapy (ACVBP or CHOP)
  Interventions: Drug: GA101; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Bleomycin; Drug: Vindesin; Drug: Vincristine
- Rituximab (Active Comparator): Rituximab - Chemotherapy (ACVBP or CHOP)
  Interventions: Drug: Rituximab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Bleomycin; Drug: Vindesin; Drug: Vincristine

INTERVENTIONS:
Drug: GA101 — in GA-ACBVP or in GA-CHOP 1000 mg on D1 and D8 (D8 in cycle 1 and 2)
  Other Names: obinutuzumab; Gazivaro
  Arms: GA101
Drug: Rituximab — in R-ACBVP or in R-CHOP 375 mg/m² on D1
  Other Names: Mabthera
  Arms: Rituximab
Drug: Doxorubicin — in ACBVP : 75 mg/m² on D1 in CHOP : 50 mg/m² on D1
Drug: Cyclophosphamide — in ACBVP : 1200 mg/m² on D1 in CHOP : 750 mg/m² on D1
Drug: Prednisone — in ACBVP : 60 mg/m² from D1 to D5 in CHOP : 40 mg/m² from D1 to D5
Drug: Bleomycin — in ACBVP 10 mg from D1 to D5
Drug: Vindesin — in ACBVP 2 mg/m² from D1 to D5
Drug: Vincristine — in CHOP 1,4 mg/m² on D1

SUMMARY:
This study is designed to investigate:

* the interest of a new monoclonal antibody (GA101)versus rituximab
* the interest of PET to identify early responders

Patients will receive either rituximab (standard treatment), either GA101 (study treatment), according to the randomization arm.

The monoclonal antibody will be associated to a chemotherapy: CHOP or ACVBP according to site's choice.A PET scan will be done before inclusion, after 2 chemotherapy cycles, and after 4 chemotherapy cycles, to identify early patients responders, for who consolidation with ASCT is not required.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20+ diffuse large B cell lymphoma (WHO Classification)
* Baseline PET scan available with at least one hypermetabolic lesion
* Aged ≥ 18 years and ≤ 60 years
* Eligible for autologous stem cell transplant
* Patient not previously treated
* Age adjusted International Prognostic Index (aa-IPI) equal to 1, 2 or 3
* Life expectancy ≥ 3 months
* Negative HIV, HBV (anti-HBc negativity) and HCV serologies before inclusion
* Having signed a written informed consent
* Having ability and willingness to comply with study protocol procedures
* Men must agree to use a barrier method of contraception during the treatment period and until 3 months after the last dose of GA101 or rituximab, or ACVBP14 or CHOP14 chemotherapy, whichever is longer
* Women of childbearing potential must agree to use an adequate method of contraception, such as oral contraceptives, intrauterine device, or barrier method of contraception during the treatment period and until 12 months after the last dose of GA101, Rituximab, ACVBP14, or CHOP14 chemotherapy, whichever is longer

Exclusion Criteria:

* Any other histological type of lymphoma
* Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included
* Central nervous system or meningeal involvement by lymphoma
* Contra-indication to any drug contained in the chemotherapy regimens
* Poor cardiac function (LVEF < 50%) on echocardiogram or MUGA scan
* Poor renal function (creatinine level > 150*mol/l or clearance < 30ml/min), poor hepatic function (total bilirubin level > 30µmol/l, transaminases > 2.5 X maximum normal level) unless these abnormalities are related to the lymphoma
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/L or platelets < 100 G/L, unless related to bone marrow infiltration
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Any serious active disease (according to the investigator's decision)
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy
* Pregnant or lactating women
* Adult patient under tutelage
* Prior history of Progressive Multifocal Leukoencephalopathy (PML)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 671 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
2-year Event Free Survival | Up to 2 years
  EFS is defined as PET positivity according to ΔSUVmax criteria after 2 or 4 induction cycles as defined by RAC (based on central PET review), progression or relapse according to Cheson 2007, modification of planned treatment out of progression or death of any cause.

SECONDARY OUTCOMES:
• Overall Response rate and Best overall response after 4 cycles and end of treatment according to Cheson 2007 criteria | Up to 3.5years
  Response will be assessed after 4 cycles and again at the end of treatment, based on RAC assessment for PET 4 and investigator assessment for EoT PET. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 2007). Overall (CR//PR) response rates and Best Response Rate will be presented. Patient without response assessment (due to whatever reason) will be considered as non-responder.
• Overall Response Rate and Best overall response after 4 cycles and end of treatment according to Cheson 1999 criteria | Up to 3.5 years
  Response will be assessed after 4 cycles and at the end of treatment, based on investigator assessment. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999). Overall (CR/CRu/PR) response rates and Best Overall Response Rate will be presented. Patient without response assessment (due to whatever reason) will be considered as non-responder.
• Duration of response (DoR) | Up to 6.5 years
  Duration of response is defined as the period from the time of attainment a CR or PR to the date of progression, relapse or death from any cause. Duration or response would be assessed as survival in the whole population, in the two inductive arms (R-Chemo14 vs GA101-Chemo14) For patients achieving a response but who have not progressed or relapsed or died at the time of analysis, DOR will be censored on the date of last disease assessment
• Progression-Free Survival (PFS) | Up to 6.5 years
  Progression-Free Survival is defined as the period from the date of randomization to the date of first documented disease progression, relapse, or death from any cause. For patients who have not progressed, relapsed, or died at the time of analysis, PFS will be censored on the date of last disease assessment. If no tumor assessments were performed after the baseline visit, PFS will be censored at the time of randomization
• Overall survival (OS) | Up to 6.5 years
  Overall survival is defined as the period from the date of randomization to the date of death from any cause. Alive patients at the time of the analysis will be censored at their last contact date
• Blood samples and on tumor tissue biopsy | Up to 6.5 years
  Analysis on blood samples and tumor tissue biopsy will be driven, in order to explore prognosis factors of the patients and their tumors that influence treatment response based on PET assessment and prognosis
• Focus on subpopulation | Up to 6.5 years
  Duration of response, PFS and OS will be performed according to treatment arms (R-Chemo14 vs GA101-Chemo14) on different analysis populations. The subpopulations are based on the outcome during the induction phase and a statistical bias could be introduced as subpopulations have not been defined at baseline.
  * Population with a Δ SUVmaxPET0-2≤66% (slow and intermediate responders),
  * Population with a Δ SUVmaxPET0-2>66% (fast responders),
  * Patients submitted to autologous stem cell transplant (PFS and OS only)
Number of stem cell collected after GA101 treatment | Up to 3.5 years
  Number of stem cell collected after GA101 administration Number of required collects to achieve 3Mcells/kg.
• Early metabolic response according to PET after 2 and 4 cycles | Up to 3.5 years
  Based on results of central PET review

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Casasnovas, MD, Study Chair — Lymphoma Study Association; Steven Le Gouill, MD, Study Chair — Lymphoma Study Association
Locations (122):
- Belgium (24):
  - ZNA Stuivenberg, Antwerp
  - Hôpital Saint Joseph, Arlon
  - RHMS Baudour, Baudour
  - AZ St Jan Brugge Oostende AV, Bruges
  - Institut Jules Bordet, Brussels
  - CHU Brugmann, Brussels
  - Hôpital Erasme, Brussels
  - Clinique universitaire Saint LUC, Brussels
  - CHU de Charleroi, Charleroi
  - Grand Hôpital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Ch Jolimont, Haine-Saint-Paul
  - AZ GROENINGE - Oncology Centre - Campus Maria's Voorzienigheid, Kortrijk
  - CHR de la Citadelle, Liège
  - CHU de Liège - Clinique Saint Joseph, Liège
  - CHU de Liège -Domaine Sart Tilman, Liège
  - CHU Ambroise Paré, Mons
  - Clinique Saint Joseph -Hôpital de Warquignies, Mons
  - Clinique Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - Heilig Hart Ziekenhuis, Roeselare
  - Centre Hospitalier de Wallonie Picarde - CHwapi, Tournai
  - CH de la Tourelle-Peltzer, Verviers
  - Université Catholique de Louvain Mont Godinne, Yvoir
- France (98):
  - CH d'Abbeville, Abbeville
  - CHU d'Amiens - Hôpital Sud, Amiens
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - CH d'Arras, Arras
  - CH d'Avignon, Avignon
  - Hôpital de Bayonne - CHU de la Côte Basque, Bayonne
  - CH de Beauvais, Beauvais
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CH de Blois, Blois
  - APHP - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH Dr Duchenne, Boulogne-sur-Mer
  - CH Fleyriat, Bourg-en-Bresse
  - CHU de Brest - Hôpital de Morvan, Brest
  - CH Brive la Gaillarde, Brive-la-Gaillarde
  - CHU de Caen, Caen
  - Centre François Baclesse, Caen
  - CH de Cannes, Cannes
  - Clinique Du Parc, Castelnau-le-Lez
  - CH de Chambéry, Chambéry
  - CHU de Châlon sur Saône, Châlon Sur Saône
  - APHP - Hôpital Antoine Béclère, Clamart
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Pôle Santé Publique, Clermont-Ferrand
  - CH de Compiègne, Compiègne
  - CH Sud Francilien, Corbeil-Essonnes
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH de Dunkerque, Dunkirk
  - Institut Daniel Hollard, Grenoble
  - CHU de Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - CH de Lens, Lens
  - CH Saint Vincent de Paul, Lille
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU Dupruytren - Limoges, Limoges
  - CH Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - CH Mantes La Jolie, Mantes-la-Jolie
  - Hôpital de la Conception, Marseille
  - Institut Paoli Calmettes, Marseille
  - CH de Meaux, Meaux
  - CH Marc Jacquet, Melun
  - Hôpital Notre Dame Bon Secours, Metz
  - CHI de Meulan, Meulan-en-Yvelines
  - CHU de Montpellier - Saint Eloi, Montpellier
  - Centre Val d'Aurélie - Paul Lamarque, Montpellier
  - Centre Auréen de Cancérologie, Mougins
  - CH de Mulhouse - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - Clinique Valdegour, Nîmes
  - CHR d'Orléans, Orléans
  - Institut Curie, Paris
  - APHP - Hôpital de la Pitié Salpetrière, Paris
  - Hôpital Cochin, Paris
  - APHP - Hôpital Necker, Paris
  - APHP - Hôpital Saint Louis, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - CH Saint Jean, Perpignan
  - CHU de Haut Lévèque, Pessac
  - Hospices Civils de Lyon - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CH d'Annecy, Pringy
  - CHU Robert Debré, Reims
  - Institut du Cancer de Courlancy, Reims
  - CHU de Rennes, Rennes
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - CH Yves Le Foll - St Brieuc, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - CHI de Poissy St Germain, Saint-Germain-en-Laye
  - Institut de Cancérologie, Saint-Priest-en-Jarez
  - CH de Saint Quentin, Saint-Quentin
  - CHU de Saint Malo, St-Malo
  - Strasbourg Oncologie Libérale, Strasbourg
  - CHU de Strasbourg, Strasbourg
  - Hopital Saint Husse, Toulon
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
  - CHU de Tours, Tours
  - CHU de Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - CH de Versailles, Versailles
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Camus V, Molina T, Desmots F, Blanc-Durand P, Kanoun S, Moslemi A, Ruminy P, Le Gouill S, Ghesquieres H, Oberic L, Morschhauser F, Tilly H, Ribrag V, Houot R, Thieblemont C, Maisonneuve H, Claves F, Bouabdallah K, Haioun C, Damaj GL, Fornecker LM, Noel R, Feugier P, Sibon D, Cartron G, Bonnet C, Bernard W, Kraeber-Bodere F, Bodet-Milin C, Jais JP, Briere J, Rossi C, Elsensohn MH, Chartier L, Itti E, Jardin F, Fest T. Interim PET after 4 cycles predicts outcome in histomolecularly confirmed primary mediastinal B-cell lymphoma. Blood Adv. 2025 May 13;9(9):2232-2246. doi: 10.1182/bloodadvances.2024015577. PMID 40030008
- [Derived] Itti E, Blanc-Durand P, Berriolo-Riedinger A, Kanoun S, Kraeber-Bodere F, Meignan M, Gat E, Gouill SL, Casasnovas RO, Bodet-Milin C. Validation of the DeltaSUVmax for Interim PET Interpretation in Diffuse Large B-Cell Lymphoma on the Basis of the GAINED Clinical Trial. J Nucl Med. 2023 Nov;64(11):1706-1711. doi: 10.2967/jnumed.123.265871. Epub 2023 Sep 21. PMID 37734837
- [Derived] Jullien M, Tessoulin B, Ghesquieres H, Oberic L, Morschhauser F, Tilly H, Ribrag V, Lamy T, Thieblemont C, Villemagne B, Gressin R, Bouabdallah K, Haioun C, Damaj G, Fornecker LM, Schiano De Colella JM, Feugier P, Hermine O, Cartron G, Bonnet C, Andre M, Bailly C, Casasnovas RO, Le Gouill S. Deep-Learning Assessed Muscular Hypodensity Independently Predicts Mortality in DLBCL Patients Younger Than 60 Years. Cancers (Basel). 2021 Sep 7;13(18):4503. doi: 10.3390/cancers13184503. PMID 34572728
- [Derived] Le Gouill S, Ghesquieres H, Oberic L, Morschhauser F, Tilly H, Ribrag V, Lamy T, Thieblemont C, Maisonneuve H, Gressin R, Bouhabdallah K, Haioun C, Damaj G, Fornecker L, Bouhabdallah R, Feugier P, Sibon D, Cartron G, Bonnet C, Andre M, Chartier L, Ruminy P, Kraeber-Bodere F, Bodet-Milin C, Berriolo-Riedinger A, Briere J, Jais JP, Molina TJ, Itti E, Casasnovas RO. Obinutuzumab vs rituximab for advanced DLBCL: a PET-guided and randomized phase 3 study by LYSA. Blood. 2021 Apr 29;137(17):2307-2320. doi: 10.1182/blood.2020008750. PMID 33211799
- [Derived] Blanc-Durand P, Jegou S, Kanoun S, Berriolo-Riedinger A, Bodet-Milin C, Kraeber-Bodere F, Carlier T, Le Gouill S, Casasnovas RO, Meignan M, Itti E. Fully automatic segmentation of diffuse large B cell lymphoma lesions on 3D FDG-PET/CT for total metabolic tumour volume prediction using a convolutional neural network. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1362-1370. doi: 10.1007/s00259-020-05080-7. Epub 2020 Oct 24. PMID 33097974